CLINICAL TRIAL: NCT04561752
Title: A Randomized, Open-Label, 2-Way Crossover, Single-Dose Food Effect Study of ZN-c5 in Healthy Adult Post-Menopausal Female Subjects
Brief Title: A Food Effect Study With ZN-c5 in Healthy Post-Menopausal Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zeno Alpha Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ZN-c5-006
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Healthy
Keywords: Randomized; Postmenopause; Female

STUDY DESIGN:
Intervention Model Description: All participants will receive the same treatment but are randomized to one of two different treatment sequences in fed and fasted states.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence A-B (Experimental): Participants will take ZN-c5 (150mg), single dose, under fasted conditions, and a week later, will take the same drug under fed conditions to determine the comparative bioavailability of ZN-c5 under these conditions.
  Interventions: Drug: ZN-c5
- Treatment Sequence B-A (Experimental): Participants will take ZN-c5 (150mg), single dose, under fed conditions, and a week later, will take the same drug under fasted conditions to determine the comparative bioavailability of ZN-c5 under these conditions.
  Interventions: Drug: ZN-c5

INTERVENTIONS:
Drug: ZN-c5 — ZN-c5 is the study drug.

SUMMARY:
This is a single-center, randomized, open-label, two-period, 2-way crossover food effect study to determine the comparative bioavailability of ZN-c5 under fed and fasting conditions, following single-dose administration of ZN-c5 capsules (150mg).

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers
* Body mass index (BMI) between > or = 18.0 kg/m2 and < or = 29.9 kg/m2, and a body weight > or = 50kg and < or = 100kg at Screening
* Non-smoker and must not have used any tobacco products within 2 months prior to Screening, or if a smoker must be currently (and for the last 2 months prior to screening) smoking < or = 2 cigarettes or equivalent per week. Current smokers must be willing to abstain from the use of tobacco and products containing nicotine from 14 days prior to administration of study drug and through the EOS visit.
* No relevant dietary restrictions, and be willing to consume a high calorie, high fat breakfast and other standard meals provided during the domiciled periods of the study
* Post-menopausal for > or = 24 months. Status will be confirmed through testing of follicle-stimulating hormone (FSH) levels > or = 40 IU/L at Screening. Participants that are post-menopausal for < or = 24 months are still potentially eligible, but will be required to have a negative serum pregnancy test result at Screening and negative urine pregnancy test result prior to study drug administration.

Exclusion Criteria:

* Any condition likely to affect the participant's ability to consume the standard meal provided during the domiciled periods of the study, or any condition that may make it difficult for the patient to comply with the requirement for fasting during the study
* Blood donation or significant blood loss within 60 days prior to the first study drug administration
* Plasma donation within 7 days prior to the first study drug administration
* Fever (body temperature > or = 38C) or symptomatic viral or bacterial infection or febrile illness within 2 weeks prior to Screening
* Positive serum pregnancy test at Screening or urine pregnancy test prior to administration of study drug (for participants who are post-menopausal for < or = 24 months only)
* Positive toxicology screening panel or alcohol breath test
* History of substance abuse or dependency or history of recreational intravenous (IV) drug use over the last 5 years (by self-declaration)
* Regular alcohol consumption within the 6 months prior to study drug administration, defined as > 21 alcohol units per week

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
AUC0-t | Days 1-4
  Area under the plasma concentration-time curve (AUC) from time zero to the last sampling time
Cmax | Days 1-4
  Maximum concentration
Tmax | Days 1-4
  Time to maximum concentration
AUC0-infinity | Days 1-4
  Area under the plasma concentration-time curve (AUC) from time zero to infinity

SECONDARY OUTCOMES:
Assess the incidence, frequency, and severity of treatment-emergent adverse events (TEAEs) | Approximately 45 days
  Safety and tolerability of ZN-c5

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Voliotis, Study Chair — Zeno Alpha Inc.
Locations (1):
- Site 1, Christchurch, New Zealand